CLINICAL TRIAL: NCT01782534
Title: Logistic Regression of Risk Factor for the 5-year Mortality of Aortic Dissection
Status: Completed | Type: Observational
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Zhishan SUN, Xiangtan City central Hospital affiliated to Central South university, Central South University
Other Study IDs: LR-RF-AD
Record Dates: First submitted 2013-01-04; First posted 2013-02-04 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Aortic Dissection
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- aortic dissection: aortic dissection

SUMMARY:
The relevant predictive hospital risk factors for 5-year mortality of patients with aortic dissection is untill unlear. The aim of this study is to collect the clinical data of 111 hospitalized patients admitted to hospital from Aug. 2001 to Aug. 2007, and statistically analyze the hospital risk factors related to 5-year mortality by univariate and multivariate binary logistic regression.

DETAILED DESCRIPTION:
Clinical data were collected from 111 hospitalized patients admitted to hospital from Aug. 2001 to Aug.2007, and the related factors for death within 5 years after the onset of dissection, which include Gender, age, history of smoking, hypertension, diabetes, renal insufficiency (azotemia), low admission diastolic blood pressure (<70mmHg), Stanford typing (Stanford A or B), long-acting calcium channel blocker treatment,ACEI /ARB treatment, endovascular stent and surgical aortic replacement,were statistically analyzed by univariate and multivariate binary logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* Stanford type A dissection
* Stanford type B dissection

Exclusion Criteria:

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: diagnosed AD patients in Our hospital From August 2001 to August2007
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2002-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
death after 5 years after the onset of dissection | 5 years
  participants have been followed for 5 years after the onset of dissection

CONTACTS AND LOCATIONS:
Overall Officials: Zhishan SUN, doctor, Principal Investigator — Central South University